CLINICAL TRIAL: NCT07310121
Title: Barriers and Enablers to Accessing Medical Care for Urinary Incontinence and Prolapse in GLobal Majority Women
Acronym: BEAM UP & GLOW
Status: Not yet recruiting | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Burdett Trust for Nursing (Other)
Responsible Party: Sponsor
Other Study IDs: B02637; 25/WA/0334 (Other: NHS Research Ethics)
Record Dates: First submitted 2025-12-02; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Pelvic Prolapse Conditions
Keywords: Pelvic organ prolapse; Pelvic floor dysfunction; Urinary incontinence
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with condition: Women with urinary incontinence or pelvic organ prolapse from an ethnic minority/global majority background who are attending a urogynaecology clinic in the Warrell Unit at Manchester University NHS Foundation Trust.
  Interventions: Other: No intervention
- Public: Women from ethnic minority/global majority background attending community groups in Greater Manchester.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
This project aims to explore barriers to treatment seeking for symptoms of prolapse and urinary incontinence in women from ethnic minority/global majority background.

This study consists of three components, each with different methodological approaches:

1. Collecting objective data using validated questionnaires Prolapse and Incontinence Knowledge Questionnaire (PIKQ), Female Genital Self-Image Scale (FGSIS-4) and prevalence and severity of urinary incontinence and pelvic organ prolapse (ICIQ-UI Short Form and ICIQ-VS), age, level of education, level of deprivation (according to postcode), faith, first or preferred language spoken, sexual orientation and employment status to explore whether these are associated with barriers to treatment seeking as measured by the Barriers to Incontinence Care Seeking Questionnaire (BICS-Q) and to estimate the prevalence of urinary incontinence and prolapse in a community group of women from an ethnic minority/global majority background
2. Collecting qualitative data via semi-structured interviews with women from an ethnic minority/global majority background who have sought treatment for urinary incontinence or pelvic organ prolapse to explore barriers they may have experienced and how these were overcome and collecting qualitative data via focus group discussions with women from an ethnic minority/global majority background who attend women's community groups
3. Zine making as a research approach is a creative, participatory method that uses the process of creating zines (small, self-published, often handmade booklets) to generate, explore, and share knowledge . Zine making blends arts-based research and participatory action research and is particularly suited for working with seldom heard communities or exploring stigmatised conditions because it gives participants creative control over how their experiences are communicated, which can be empowering, especially for individuals who are under or misrepresented in mainstream narratives . Zine making is also more accessible for individuals who do not speak English as their first or preferred language, or, have other communication barriers .

ELIGIBILITY:
Women who have been referred to MFT for the specified condition.

Inclusion Criteria:

* To be willing and able to give informed consent
* To have been born female and to currently identify as female
* To be over the age of 18 years
* To have accessed medical care for urinary incontinence or pelvic organ prolapse
* To be from an ethnic minority/ global majority background
* To be able to speak and understand English

Exclusion Criteria:

-

Women attending select community centres in Greater Manchester area.

Inclusion Criteria:

* To be willing and able to give informed consent
* To have been born female and to currently identify as a woman
* To be over the age of 18 years
* To be from an ethnic minority/ global majority background
* To be able to speak and understand either English, or a language which the community group translator can communicate in

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who have been referred to MFT for the specified condition. Women attending select community centres in Greater Manchester area.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Prolapse and Incontinence Knowledge Questionnaire (PIKQ) | 12 months
  * 24 statements, with three responses: "Agree," "Disagree," or "I don't know". Each correct answer is scored 1, incorrect or not known answers score as a 0. Total score is calculated by adding each score together with a maximum total of 24.
  * The higher the score the greater the knowledge of prolapse and incontinence.
Barriers to Incontinence Care Seeking questionnaire (BICS-Q) | 12 months
  * BICS-Q consists of 14 questions that address different barriers to incontinence care seeking.
  * Each question is scored between 0-3 based on level of agreement with the statement.
  * BICS-Q is scored on a scale of 0 to 42.
  * The higher the score the more barriers to care seeking.

SECONDARY OUTCOMES:
International Consultation on Incontinence Questionnaire (ICIQ UI Short Form) | 12 months
  * ICIQ-UI SF is scored on a scale of 0 to 21.
  * The higher the score the more severe the urinary incontinence.
International Consultation on Incontinence Questionnaire and Vaginal Symptoms (ICIQ VS) | 12 months
  * ICIQ-VS is scored on a scale of 0 to 53.
  * The higher the score the more severe the vaginal symptoms.
Female Genital Self-Image Scale (FGSIS-4) | 12 months
  * FGSIS-4 is scored on a scale of 4-16.
  * The higher the score the greater the female genital self-image.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Dwyer, PhD, Principal Investigator — Manchester University Hospitals NHS Foundation Trust
Locations (1):
- Manchester University Hospitals NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No